CLINICAL TRIAL: NCT06940804
Title: Open-label Phase II Trial to Evaluate Anti-tumor Activity and Safety of CLDN6 CAR-T ± CLDN6 RNA-LPX in Male Participants With Relapsed or Refractory Claudin 6-positive Testicular or Extragonadal Germ Cell Tumors
Brief Title: A Clinical Study Investigating the Therapeutic Effects and Safety of an Investigational Cell Therapy Given With and Without an Additional Investigational Product in Males With Testicular Cancer or a Form of Cancer That Developed From Sperm
Acronym: AVENTURINE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT211-02; 2024-511941-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Testicular Germ Cell Tumor; Extragonadal Germ Cell Tumor
Keywords: Advanced germ cell tumor; Metastatic germ cell tumors; CLDN6-positive relapsed or refractory advanced solid tumors; Salvage therapy; Testicular cancer; Immunotherapy; Autologous T-cells
MeSH Terms: conditions — Testicular Germ Cell Tumor; Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Lead-in Part - CLDN6 CAR-T (dose level 1) + CLDN6 RNA-LPX (Experimental)
  Interventions: Biological: CLDN6 CAR-T; Biological: CLDN6 RNA-LPX
- Safety Lead-in Part - CLDN6 CAR-T (dose level 2) (Experimental)
  Interventions: Biological: CLDN6 CAR-T
- Safety Lead-in Part - CLDN6 CAR-T (dose level 2) + CLDN6 RNA-LPX (Experimental)
  Interventions: Biological: CLDN6 CAR-T; Biological: CLDN6 RNA-LPX
- Main Part - Selected dose of CLDN6 CAR-T + CLDN6 RNA-LPX (Experimental): Doses as selected from the Safety Lead-in Part
  Interventions: Biological: CLDN6 CAR-T; Biological: CLDN6 RNA-LPX

INTERVENTIONS:
Biological: CLDN6 CAR-T — Intravenous (IV) infusion
Biological: CLDN6 RNA-LPX — IV injection
  Arms: Main Part - Selected dose of CLDN6 CAR-T + CLDN6 RNA-LPX; Safety Lead-in Part - CLDN6 CAR-T (dose level 1) + CLDN6 RNA-LPX; Safety Lead-in Part - CLDN6 CAR-T (dose level 2) + CLDN6 RNA-LPX

SUMMARY:
This study is designed to evaluate the safety, efficacy, cellular kinetics, and immunogenicity of Claudin 6 (CLDN6) Chimeric antigen receptor T cell (CAR-T) ± CLDN6 ribonucleic acid-lipoplex (RNA-LPX) in participants born male with relapsed or refractory CLDN6-positive testicular or extragonadal germ cell tumors (GCTs) after prior salvage therapy.

DETAILED DESCRIPTION:
The study will consist of two parts. The Safety Lead-in Part will evaluate safety and tolerability of CLDN6 CAR T ± CLDN6 RNA-LPX therapy in three arms with different dosing regimens. In the Safety Lead-in Part, participants will be randomized in a 1:1:1 ratio. Data from the Safety Lead-in Part up to the cut off will be used to select the dose for the single-arm Main Part of the study.

To increase the potency of the transferred CAR-T cells, a lymphodepleting chemotherapy regimen (comprising fludarabine and cyclophosphamide) will be administered in participants prior to infusion of CLDN6 CAR-T.

It is expected that it will take approximately 28 months for each participant to complete screening, apheresis, pre-treatment, treatment, and primary follow-up.

Participants who receive a CLDN6 CAR-T infusion will complete the long-term follow-up (LTFU) to assess safety and efficacy of the CLDN6 CAR-T treatment for a total of 15 years after CLDN6 CAR-T infusion. No investigational medicinal product (IMP) will be administered during the LTFU.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a histologically confirmed diagnosis of a testicular or extragonadal GCT of extracranial origin.
* Evidence of measurable disease by RECIST 1.1 or if RECIST 1.1 evaluation is not possible, elevation of serum tumor marker(s) (AFP or βhCG).
* Participants with evidence of progressive or recurrent metastatic GCT defined as meeting at least one of the following criteria:

  * Tumor biopsy of new or growing or unresectable lesions demonstrating viable non-teratomatous GCT. In the event of an incomplete gross resection where viable GCT is found, participants will be considered eligible for this study.
  * Elevated serum tumor markers (AFP or ßhCG) that are increasing. Increase of an elevated lactate dehydrogenase alone does not constitute progressive disease.
  * Development of new or enlarging lesions in the setting of persistently elevated AFP or ßhCG, even if the markers are not continuing to rise.
* Participants must have received prior high-dose chemotherapy with autologous stem cell transplantation or conventional dose chemotherapy as salvage therapy. There is no maximum limit for the number of prior treatments.
* Have a CLDN6-positive tumor assessed using an analytically validated immunohistochemistry assay at a central laboratory.
* Have an Eastern Cooperative Oncology Group performance status of 0 to 1.
* Have laboratory tests of adequate organ function as defined in the protocol.

Key Exclusion Criteria:

* Had major surgery within the 4 weeks before the first dose of study treatment.
* Have received a prior CLDN6 CAR-T therapy.
* Are receiving systemic (oral or IV) steroid therapy >10 mg prednisolone daily, or its equivalent, for an underlying condition.
* Have unresolved side effects of any prior therapy or procedures not recovered to CTCAE version 5.0 Grade 1 or lower, except for AEs not constituting a safety risk by investigator judgment.
* Have a pure teratoma, or pure teratoma with somatic-type malignancy or a combination of these histologies without any additional histologic subtype.
* Have current evidence of active and/or uncontrolled brain or spinal metastases.
* Have an active autoimmune disease or any active immunologic disorder requiring immunosuppression with steroids or other immunosuppressive agents (protocol-defined exceptions apply). Note: Participants may be included if their disease is well controlled without the use of immunosuppressive agents, at the discretion of the investigator.
* Have a history of another primary cancer within the 24 months prior to signing the main informed consent form (exceptions for definitely treated malignancies that have been in complete remission for more than 24 months apply).
* Receipt of allogeneic stem cell transplantation in the 5 years prior to study enrollment.
* Have cardiac conditions defined as exclusionary per protocol.
* Have any concurrent conditions that could pose an undue medical hazard or interfere with the interpretation of the study results.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2042-06 (Estimated); Study Completion 2042-06 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-in Part: Occurrence of treatment emergent adverse events (TEAEs) including Grade ≥3, adverse events of special interest (AESIs) and serious or fatal TEAEs by casual relationship to study treatment | Up to 110 weeks after first dose of IMP
  For each treatment arm
Main Part: Overall response rate (ORR) assessed by the blinded independent central review (BICR) | Up to 110 weeks after first dose of IMP
  Defined as the percentage of participants in whom a confirmed complete response (CR) or partial response (PR) (per response evaluation criteria in solid tumors version 1.1 ([RECIST 1.1]) is observed as best overall response
LTFU: Occurrence of AEs suspected to be related to CLDN6 CAR-T | Up to 15 years after CLDN6 CAR-T administration
  AEs may include: new malignancy (hematologic or solid) from genetically modified cells; new neurologic disorder, or exacerbation of a pre-existing disorder; new rheumatologic or autoimmune disorder, or exacerbation of a prior rheumatologic or other autoimmune disorder; new hematologic disorder; other new clinical condition considered by the investigator to be related to the prior genetically engineered T-cell therapy.

SECONDARY OUTCOMES:
Safety Lead-in and Main Part: Occurrence of TEAEs including Grade ≥3, AESIs, and serious or fatal TEAEs by casual relationship to study treatment | From first dose of IMP until 90 days after last dose of IMP, or until a new anticancer therapy is started, whichever occurs first
  For each treatment arm
Safety Lead-in and Main Part: Geometric mean of pharmacokinetic parameter maximum concentration (Cmax) of CLND6 CAR-T | Up to 97 weeks after first IMP dose
  For each treatment arm using CLND6 CAR-T concentration in blood
Main Part: Geometric mean of pharmacokinetic parameter Cmax of interleukin (IL)-6 | Up to 97 weeks after first IMP dose
  From baseline until last available sample
Safety Lead-in and Main Part: Geometric mean of pharmacokinetic parameter time to maximum concentration (Tmax) of CLND6 CAR-T | Up to 97 weeks after first IMP dose
  For each treatment arm using CLND6 CAR-T concentration in blood
Main Part: Geometric mean of pharmacokinetic parameter Tmax of IL-6 | Up to 97 weeks after first IMP dose
  From baseline until last available sample
Safety Lead-in and Main Part: Geometric mean of pharmacokinetic parameter area under the time concentration curve (AUC) of CLND6 CAR-T | Up to 97 weeks after first IMP dose
  For each treatment arm using CLND6 CAR-T concentration in blood
Safety Lead-in and Main Part: Overall response rate (ORR) assessed by the investigator | Up to 110 weeks after first dose of IMP
  Defined as the percentage of participants in whom a confirmed complete response (CR) or partial response (PR) is observed as best overall response. Tumor response will be assessed by the investigator per RECIST 1.1. In the Safety Lead-in Part, tumor assessment will also be made based on reduction of the serum tumor marker(s) (alpha fetoprotein [AFP]/beta human chorionic gonadotropin [βhCG]).
Safety Lead-in and Main Part: Disease control rate (DCR) assessed by the investigator | Up to 110 weeks after first dose of IMP
  Defined as the percentage of participants in whom a CR, PR, or stable disease (SD) is observed as best overall response. Tumor response will be assessed per RECIST 1.1. In the Safety Lead-in Part, tumor assessment will also be made based on reduction of the serum tumor marker(s) (alpha fetoprotein [AFP]/beta human chorionic gonadotropin [βhCG]).
Main Part: DCR assessed by BICR | Up to 110 weeks after first dose of IMP
  Defined as the percentage of participants in whom a CR, PR, or SD is observed as best overall response. Tumor response will be assessed per RECIST 1.1
Main Part: Progression-free survival (PFS) assessed by the investigator | Up to 110 weeks after first dose of IMP
  Defined as the time from first dose of CLDN6 CAR-T to progressive disease (PD) or death from any cause, whichever occurs first. Tumor response will be assessed per RECIST 1.1
Main Part: PFS assessed by BICR | Up to 110 weeks after first dose of IMP
  Defined as the time from first dose of CLDN6 CAR-T to PD or death from any cause, whichever occurs first. Tumor response will be assessed per RECIST 1.1
LTFU: PFS assessed by the investigator | Up to 15 years after the last IMP administration
  Defined as the time from first dose of CLDN6 CAR-T to first objective progressive disease per RECIST 1.1 and/or based on reduction of the serum tumor marker(s) (AFP/βhCG), or death from any cause, whichever occurs first.
Main Part: Duration of response (DOR) assessed by the investigator | Up to 110 weeks after first dose of IMP
  Defined as the time from first objective response (CR or PR) to first occurrence of tumor progression, or death from any cause, whichever occurs first. Tumor response will be assessed per RECIST 1.1.
Main Part: DOR assessed by BICR | Up to 110 weeks after first dose of IMP
  Defined as the time from first objective response (CR or PR) to first occurrence of tumor progression, or death from any cause, whichever occurs first. Tumor response will be assessed per RECIST 1.1.
Main Part: Overall survival (OS) | Up to 97 weeks after first dose of IMP or until death, whichever occurs first
  Defined as the time from first dose of CLDN6 CAR-T to death from any cause
LTFU: OS | Up to 15 years from last genetically engineered T-cell infusion or until death, whichever occurs first
  Defined as the time from first dose of CLDN6 CAR-T to death from any cause
Main Part: Percentage of participants with pre-existing anti-chimeric antigen receptor (CAR) antibodies prior to CLDN6 CAR-T infusion | On Day 1 prior to CAR-T infusion
  For each treatment arm using CLND6 CAR-T concentration in blood and of IL-6 from baseline until last available sample
Main Part: Percentage of participants with treatment-emergent anti-CAR antibodies post-CLDN6 CAR-T infusion until last available sample | Up to 97 weeks after first dose of IMP
  Anti-CAR antibodies including both treatment-induced and treatment-boosted

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE

IPD SHARING:
Plan to Share IPD: No